CLINICAL TRIAL: NCT05737329
Title: Optimization of Management Tactics for Women With Premature Ovarian Insufficiency, Taking Into Account Their Clinical and Hormonal Profile
Brief Title: Efficacy, Safety, and Tolerability of Higher Doses Estrogen Therapy in Women With Premature Ovarian Insufficiency
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: №2-07/02.2019
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Primary Ovarian Insufficiency
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Intervention Model Description: Women with POI taking standard-dose estradiol hormone replacement therapy (E2/dydrogesterone (oral) (2.0/10 mg)) were invited to the study. We conducted a pilot study designed to compare the effectiveness of oral estradiol (2mg/ day) and Transdermal estradiol gel 0.1% (Gel sachet 1.0mg/ day) as standard-dose estradiol hormone replacement therapy. The obtained results on the absence of a significant difference in the effect of the above therapy made it possible to justify the prescription of higher doses of estrogens without prior switching from oral to transdermal therapy in equivalent doses in all study participants. Study participants will consistently receive Transdermal estradiol gel 0.1% (Gel sachet 1.5mg/ day) and Transdermal estradiol gel 0.1% (Gel sachet 2.0mg/ day) (both with 200mg micronized progesterone administered vaginally for 14days per cycle) with an outcome assessment at each stage of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transdermal estradiol gel 0.1% 1.5mg/ day (Other): Patient will be given Hormone Replacement Therapy (HRT) in the form of: Transdermal estradiol gel 0.1% 1.5mg (Gel sachet) in continuous daily regimen. The progesterone component of HRT (200mg micronized progesterone administered vaginally) will be given for 14 days, starting from day 14 through day 28 of each cycle.
  Interventions: Drug: Transdermal estradiol gel 0.1% 1.5mg/ day; Drug: Transdermal estradiol gel 0.1% 2.0mg/ day
- Transdermal estradiol gel 0.1% 2.0mg/ day (Other): Patient with insufficient effect from previous treatment estradiol gel 0.1% 1.5mg will be given HRT in the form of: Transdermal estradiol gel 0.1% 2.0mg (Gel sachet) in continuous daily regimen. The progesterone component of HRT (200mg micronized progesterone administered vaginally) will be given for 14 days, starting from day 14 through day 28 of each cycle.
  Interventions: Drug: Transdermal estradiol gel 0.1% 1.5mg/ day; Drug: Transdermal estradiol gel 0.1% 2.0mg/ day

INTERVENTIONS:
Drug: Transdermal estradiol gel 0.1% 1.5mg/ day — Estradiol gel 0.1% 1.5mg/ daily + Micronized Progesterone 200mg
Drug: Transdermal estradiol gel 0.1% 2.0mg/ day — Estradiol gel 0.1% 2.0mg/ daily + Micronized Progesterone 200mg

SUMMARY:
The goal of this study is to assess the effects of higher doses versus standard hormone therapy on quality of life (QoL), symptoms due to estrogen deficiency, and bone health in women with premature ovarian insufficiency (POI).

The efficacy of the hormonal treatment will be assessed clinically and also by measuring serum concentrations of Estradiol (E2), Follicle-Stimulating Hormone (FSH), Luteinizing hormone (LH), total Testosterone (T), Estrone (E1), E1 sulfate (E1S), and Sex Hormone Binding Globulin (SHBG). Bone mineral density (BMD) will be measured using dual-energy X-ray absorptiometry. Safety will be assessed by measuring endometrial thickness with Gynecological transvaginal ultrasound (TVS), treatment-related adverse events (AEs) and treatment-emergent AEs monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients with karyotypically normal spontaneous POI diagnosed before the age of 40. POI as defined by: change in menstrual function (oligomenorrhea and/or amenorrhea for at least 4 months), elevated serum follicle stimulating hormone (FSH ≥ 25 IU/L with 4 to 6 weeks interval)
* Between 18-45 years of age
* Use of standard-dose estradiol HRT (Estradiol 2 mg+ Dydrogesterone10 mg) for at least the last 12 months
* Signed informed consent before inclusion in the study

Exclusion Criteria:

* Any contraindication to HRT per the current drug labels. These could include, but are not limited to: history of venous thromboembolism, estrogen-sensitive cancer history, regular cigarette smoking and history of or active liver disease, bleeding from the genital tract of unknown origin, etc.
* POI due to cytotoxic chemotherapy or radiation therapy, surgery
* Diseases that may be associated with hot flashes (such as pheochromocytoma, hyperthyroidism, medullary carcinoma of the thyroid, acromegaly, pancreatic islet-cell tumors, renal cell carcinoma, carcinoid syndrome, systemic mast cell disease, neurological flushing, emotional flushing, spinal cord injury)
* Taking medications that can also cause hot flashes (such as Tamoxifen, Raloxifene, Tricyclic antidepressants, Monoamine oxidase inhibitors, Calcium channel blockers, Depo leuprolide, Clomiphene, Serotonin uptake inhibitors)
* Severe somatic conditions (uncontrolled hypertension, kidney disease, liver disease, etc.)
* Diseases with impaired thyroid and adrenal gland function
* Refusal to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the severity of estrogen deficiency symptoms | 3 months
  The Green scale questionnaire was used initially and after 3 months against the background of HRT. The questionnaire includes 21 questions from 0 to 3 points, where a lower score means a better result.
Changing the assessment of quality of life using the Short Form Health Survey-36 (SF-36) | 3 months
  The SF-36 is a generic QoL instrument. It consists of 36 items organized into eight domains: Physical Function (AF), Physical Role Function (RF), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Function (SF), Emotional Role Function (RE), and Mental Health (SM) as well as an item on the change of General Health. The scores of each domain have been converted into a scale from 0 to 100. Lower scores are indicative of worse conditions.
Changing the assessment of menopause-related quality of life measured using the Menopause-Specific Quality of Life (MENQOL) questionnaire. | 3 months
  The MENQOL questionnaire is a self-administered instrument. This validated questionnaire (range 1-8) assesses four quality of life domains; physical (16 items), vasomotor (3 items), psychosocial (7 items) and sexual (3 items). Scoring generates 4 domain scores and a total score, the mean of the 4 domain scores. Identical scoring for each of the four MENQOL domains is used. A "0" is identical that the woman has not experienced this specific symptom in the previous month; Score "1" demonstrates that the woman experienced the symptom, but it did not bother her; Scores "2" through "7" demonstrate an increasing level of the bothering symptom, so that these scores indicate increasing levels of bother experienced from the symptom and correspond to the ''1'' through ''6'' checkboxes on the MENQOL. With increasing MENQOL scores, levels of bother experienced from the symptom are increased as well.

SECONDARY OUTCOMES:
Сhanges in the level of sex hormones after using higher doses estrogen therapy | Assessment of changes in the level of sex hormone in peripheral blood: testosterone (nmol/l). Reference values: 0,52 - 2,5 nmol/l. Blood sampling is performed at baseline and after 3 months.
  Assessment of changes in the level of sex hormone in peripheral blood: estradiol (pmol/l). Reference values: 150 - 450 pmol/l. Blood sampling is performed at baseline and after 3 months.
Сhanges in the level of sex hormones after using higher doses estrogen therapy | 3 months
  Assessment of changes in the level of sex hormone in peripheral blood: total testosterone (nmol/l). Reference values: 0,52 - 2,5 nmol/l. Blood sampling is performed at baseline and after 3 months.
Сhanges in the level of FSH after using higher doses estrogen therapy | 3 months
Сhanges in the level of E1 after using higher doses estrogen therapy | 3 months
Сhanges in the level of E1S after using higher doses estrogen therapy | 3 months
Сhanges in the level of SHBG after using higher doses estrogen therapy | 3 months
Bone mineral density (BMD) response to using higher doses estrogen therapy for 12 Months | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Averkova, Study Chair — FSBI "National Medical Research Center for Obstetrics, Gynecology and Perinatology named after Academician V.I.Kulakov" Ministry of Healthcare of the Russian Federation
Locations (1):
- Federal State Budget Institution Research Center for Obstetrics, Gynecology and Perinatology Ministry of Healthcare, Moscow, Russia